CLINICAL TRIAL: NCT03172247
Title: How Diabetic Patient Are Taken Care in Cardiology Service Actually?
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CARDIABET
Record Dates: First submitted 2017-05-24; First posted 2017-06-01 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Diabetes
Keywords: cardiology diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Care of the diabetes is multidisciplinary with the involvment either private and hospital specialist

ELIGIBILITY:
Inclusion Criteria:

* evey patient admitted in cardiology department more than 24 hours
* 18 years old and above
* accepted to participate
* patient treated by insuline and/or with oral antidiabetic treatment
* Type 2 diabetes

Exclusion Criteria:

* Type 1 diabetes
* patient admitted for angiography
* iatrogenic hyperglycaemia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We select every day patient admitted in cardiology department with antidiabetic treatment
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Combined endpoint of diabetic hospitalized patients | During hospitalization
  Combined endpoint are glycemia dosage, glycosylated hémoglobin,insulinotherapy,

IPD SHARING:
Plan to Share IPD: No